CLINICAL TRIAL: NCT05420740
Title: Impact of Aerobika® Oscillating Positive Expiratory Pressure (OPEP) in Improving Small Airway Disease and COPD Assessment Test (CAT) Score in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Impact of Aerobika OPEP in Improving Small Airway Parameters in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FF-2021-175
Record Dates: First submitted 2022-05-09; First posted 2022-06-15 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: COPD
Keywords: COPD; Small airway disease; Impulse Oscillometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD patients with Small Airway Disease (Experimental): Subjects will be given Aerobika OPEP and IOS, CAT score, Spirometry, 6MWT and Exacerbation were assessed at Week 0, Week 12 and Week 24
  Interventions: Device: Aerobika OPEP

INTERVENTIONS:
Device: Aerobika OPEP — Subjects given Aerobika OEP to assess changes in small airway disease parameter , CAT Score , 6 minute walking test and exacerbation

SUMMARY:
Research Background Chronic obstructive pulmonary disease (COPD) is a progressive chronic lung disease that makes breathing difficult with mucus build-up in the inflamed airway and lungs hyperinflation due to expiratory flow limitation. Global Initiative for Chronic Obstructive Lung Disease (GOLD) defines COPD as a common, preventable and treatable disease with significant morbidity and mortality, and incurs intensive expenditure of healthcare resources. This disease is currently the fourth leading cause of death in the world but is projected to be the 3rd leading cause of death by 2020. In 2012, global death from COPD accounted about 6% which equal to more than 3 million deaths in world population. The mortality burden of COPD is expected to rise to 8.6% by 2030. In Malaysia, the prevalence of moderate to severe COPD in Malaysia in 2010 is 4.7% which equals to 448,000 cases.

COPD is attributed by long-term exposure to noxious particles and toxic gases. Tobacco smoking is the main cause of COPD globally. The Third National Health and Morbidity Survey (NHMS III) conducted in Malaysia in 2006 showed that the prevalence of male ever smokers was 57.6% and in female is 2.5%. Other than that, inhalation of organic or chemical dust and fumes, and biomass exposure also among the risk factors of COPD. Exposure to noxious particles will cause activation of inflammatory immune responses. However, continuous and repetitive exposure towards these noxious particles will lead to tissue remodelling in small airways causing smooth muscle hypertrophy and fibrosis causing major site of obstruction in COPD.

In COPD patients, the small airways represent the key sites of airflow obstruction, and small airway disease (SAD) is considered a functional hallmark of disease. The presence of SAD progressively increases with higher GOLD classifications and it is closely related to the high impact of disease measured by COPD Assessment Test (CAT) questionnaire. Distributions of SAD among COPD patients classified according to GOLD classification. In each of GOLD A, B, C and D class, the prevalence of SAD are 49%, 88%, 61%, and 96% respectively. As presence of SAD is closely related to high impact of disease with CAT score ≥10 , they tend to have more symptoms.

DETAILED DESCRIPTION:
IOS is a simple, non-invasive method requiring only passive patient cooperation without special manoeuvre for evaluation of lung function through the measurement of both airway resistance and airway reactance. The pressure-flow oscillations are applied at the mouth superimposed on the subject's tidal breaths to measure respiratory system resistance and reactance at different oscillation frequencies. It uses sound waves to rapidly detect airway changes. When analysed, these pressure signals separately quantify the degree of obstruction in the central and peripheral airways. In IOS, it enables measurement of total respiratory resistance (R5) and proximal respiratory resistance (R20), with the R5-R20 difference reflecting small airway resistance. Small airway disease is significance if R5-R20 > 0.71 cmH2O/L/sec.

Treatment of COPD requires combination of pharmacological and non-pharmacological approaches. In non-pharmacological treatment, chest physiotherapy and pulmonary rehabilitation is the cornerstone of management of COPD patients. It can result in improvement of symptoms, increased exercise capacity, and improvement in lung functions. By early detection of SAD in COPD, it enables the physician to offer patients with a more targeted approach therapy, for example the use of small particle size inhalers or mechanical intervention for example oscillating positive expiratory device (OPEP), such as Aerobika®.

ELIGIBILITY:
Inclusion criteria:

* Age 40 years or older
* COPD diagnosed according to the GOLD guidelines: GOLD 2 - GOLD 4
* Stable COPD patients with mucus hyperproduction: coughed and brought up sputum "several days a week" (>2 days a week) or "almost every day" in the month prior to the study
* Patients who can perform IOS
* Patients who can perform spirometry
* Patients who can perform 6MWT

Exclusion Criteria:

* COPD diagnosed according to the GOLD guidelines: GOLD 1
* Diagnosis of other chronic lung diseases: Asthma, Asthma-COPD Overlap, Interstitial Lung Disease, Bronchiectasis, Lung Cancer
* Patients with contraindication for spirometry: recent cardiac complications, major surgery, severe advanced respiratory disease, or those with cognitively or neurologically impairment
* Patients not recommended for OPEP: neuromuscular weakness, recent facial, oral or skull surgery or trauma, recent oesophageal surgery, active haemoptysis, acute sinusitis, untreated pneumothorax, known or suspected tympanic membrane rupture or other middle ear pathology, overt right-sided heart failure
* Patients with contraindication for 6 minute walking test
* Patient unable or unwilling to give informed consent
* Change of inhaler during study period

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate change of small airway parameter using impulse oscillometry after introduction of Aerobika® OPEP among COPD patients . | 3 months and 6 months
  Comparing change of small airway parameters using impulse oscillometry pre and post introduction of Aerobika OPEP; Parameters used are R5, R5-R20, X5,AX

SECONDARY OUTCOMES:
To evaluate change of CAT score | 3 and 6 months.
  Comparing change of CAT Score using questionairre pre and post introduction of Aerobika OPEP. Cat Score range 0-40 (0-not affected by symptoms, 40 marked affected by symptoms)
To evaluate changes of lung function (using spirometry) | 3 and 6 months.
  Comparing changes of lung function (FEV1 %) pre and p ost introduction of Aerobika OPEP
To evaluate changes of exercise capacity in metres (using 6-minute walking test) | 3 and 6 months.
  Comparing changes of exercise capacity in metres (using 6-minute walking test) OPEP
To evaluate moderate and severe exacerbation rates after Aerobika® OPEP device usage | 3 and 6 months.
  Comparing frequency of exacerbation (number of events ) and number of hospital admissions

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cost-effectiveness of the Aerobika* oscillating positive expiratory pressure device in the management of COPD exacerbations. Int J Chron Obstruct Pulmon Dis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5655131/
- See also: Economic Burden of Chronic Obstructive Pulmonary Disease Patients in Malaysia: A Longitudinal Study — https://link.springer.com/article/10.1007/s41669-020-00214-x
- See also: Significances of spirometry and impulse oscillometry for detecting small airway disorders assessed with endobronchial optical coherence tomography in COPD — http://doi.org/10.2147/COPD.S172639
- See also: Small Airway Disease in Asthma and COPD: Clinical Implications — https://doi.org/10.1378/chest.10-1210

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT05420740/Prot_SAP_ICF_000.pdf